CLINICAL TRIAL: NCT01835158
Title: Randomized Phase II Study Comparing Cabozantinib (NSC #761968) With Commercially Supplied Sunitinib in Patients With Previously Untreated Locally Advanced or Metastatic Renal Cell Carcinoma
Brief Title: Cabozantinib-s-malate or Sunitinib Malate in Treating Patients With Previously Untreated Locally Advanced or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00820; NCI-2013-00820 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A031203; A031203 (Other: Alliance for Clinical Trials in Oncology); A031203 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-12

CONDITIONS: Clear Cell Renal Cell Carcinoma; Metastatic Kidney Carcinoma; Stage III Renal Cell Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (cabozantinib-s-malate) (Active Comparator): Patients receive cabozantinib-s-malate PO QD for 6 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis
- Arm II (sunitinib malate) (Active Comparator): Patients receive sunitinib malate PO QD for 4 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL-184; XL184
  Arms: Arm I (cabozantinib-s-malate)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent
  Arms: Arm II (sunitinib malate)

SUMMARY:
This randomized phase II trial studies how well cabozantinib-s-malate works compared to sunitinib malate in treating patients with previously untreated kidney cancer that has spread from where it started to nearby tissue or lymph nodes or to other places in the body. Cabozantinib-s-malate and sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether cabozantinib-s-malate is more effective than sunitinib malate in treating patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if patients with renal cancer treated with cabozantinib (cabozantinib-s-malate) will have improved progression-free survival compared to patients treated with sunitinib (sunitinib malate).

SECONDARY OBJECTIVES:

I. To determine whether the response rate of patients with renal cancer treated with cabozantinib will be higher when compared with patients treated with sunitinib.

II. To determine whether patients with renal cancer treated with cabozantinib will have an improved overall survival when compared with patients treated with sunitinib.

TERTIARY OBJECTIVES:

I. To determine whether renal cancer patients with high MET expression by immunohistochemistry (IHC) have improvement in progression-free survival compared to patients with low MET expression on both arms of this study.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cabozantinib-s-malate orally (PO) once daily (QD) for 6 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive sunitinib malate PO QD for 4 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Renal cell carcinoma with some component of clear cell histology; histologic documentation of metastatic disease is not required
* Locally advanced (defined as disease not amenable to curative surgery or radiation therapy) or metastatic renal cell carcinoma (RCC) (equivalent to stage IV RCC, according to American Joint Committee on Cancer [AJCC] staging)
* Eligible patients must be intermediate/poor risk, per the International Metastatic Renal Cell Carcinoma (mRCC) Database Consortium (Heng) criteria; patients must therefore have as one or more of the following six factors:

  * Time from diagnosis of RCC to systemic treatment < 1 year

    * Note: systemic treatment refers to the initiation of A031203 protocol treatment
  * Hemoglobin < the lower limit of normal (LLN)
  * Corrected calcium > the upper limit of normal (ULN)
  * Karnofsky performance status < 80%
  * Neutrophil count > ULN
  * Platelet count > ULN
* No radiographic evidence of cavitating pulmonary lesion(s)
* No tumor invading the inferior vena cava (IVC) or superior vena cava (SVC) blood vessels
* No evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days prior to registration
* No prior systemic treatment for RCC; supportive therapies such as bisphosphonates (zoledronic acid) or denosumab are permitted
* Patients must not have had a major surgical procedure or significant traumatic injury within 6 weeks prior to study registration, and must have fully recovered from any such procedure; however, patients who have had a nephrectomy may be enrolled 4 weeks after surgery, providing there are no wound-healing complications; the following are not considered to be major procedures: thoracentesis, paracentesis, port placement, laparoscopy, thoracoscopy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, incisional biopsies, imaging-guided biopsy for diagnostic purposes, and routine dental procedures
* Radiation:

  * To the brain, thoracic cavity, abdomen, or pelvis must be completed at least 90 days before registration;
  * To bone must be completed at least 14 days before registration; and
  * To any other sites must be completed at least 28 days before registration In all cases, there must be complete recovery and no ongoing complications from prior radiation therapy
* No chronic concomitant treatment of strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers or inhibitors; patients may not have received a strong CYP3A4 inducer within 12 days prior to registration nor a strong CYP3A4 inhibitor within 7 days prior to registration
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria; lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2 cm with conventional techniques or as >= 1 cm with spiral computed tomography (CT) scan
* No active brain metastases; patients with treated, stable brain metastases for at least three months are eligible as long as they meet the following criteria:

  * Treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 3 months, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or CT); (stable dose of anticonvulsants are allowed); treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, linear accelerator [LINAC], or equivalent) or a combination as deemed appropriate by the treating physician; patients with central nervous system (CNS) metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to registration are not eligible
  * Baseline brain imaging (MRI/CT) is required
* No serious non-healing wound, ulcer, or bone fracture requiring intervention within 28 days prior to registration
* No arterial thrombotic events within 6 months prior to registration, including transient ischemic attack (TIA), cerebrovascular accident (CVA), peripheral arterial thrombus, unstable angina or angina requiring surgical or medical intervention in the 6 months prior to registration, or myocardial infarction (MI); patients with clinically significant peripheral artery disease (i.e., claudication on less than one block), significant vascular disease (i.e., aortic aneurysm, history of aortic dissection), or any other arterial thrombotic event are ineligible
* No history of pulmonary embolism or untreated deep venous thrombosis (DVT) within 6 months prior to registration; note: patients with recent DVT who have been treated with therapeutic anticoagulation with low molecular weight heparin for at least 6 weeks are eligible; patients receiving therapeutic warfarin (> 2 mg/day) are not eligible; patients on warfarin may be switched to low molecular weight heparin at the discretion of the treating physician
* No inadequately controlled hypertension (defined as a blood pressure of >= 150 mmHg systolic and/or >= 90 mmHg diastolic), or any prior history of hypertensive crisis or hypertensive encephalopathy
* No New York Heart Association (NYHA) class >= 2 congestive heart failure
* Ejection fraction on echocardiogram (Echo) or multi gated acquisition scan (MUGA) > 50%
* No corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before randomization; note: if initial QTcF is found to be > 500 ms, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed; if the average of these three consecutive results for QTcF is =< 500 ms, the subject meets eligibility in this regard
* No history of congenital QT syndrome
* No unstable cardiac arrhythmia within 6 months prior to registration
* No evidence of any of the following:

  * Clinically-significant gastrointestinal bleeding within 6 months before registration; or
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months before registration; or
  * Any other signs indicative of pulmonary hemorrhage within 3 months before registration
* No history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, bowel obstruction, or gastric outlet obstruction within 6 months prior to registration and complete healing/resolution prior to registration; no percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months prior to registration
* No active peptic ulcer disease, within 28 days before registration
* No inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis within 28 days before registration
* No malabsorption syndrome within 28 days before registration
* No uncompensated hypothyroidism; patients with hypothyroidism on therapy are required to have thyroid stimulating hormone (TSH) within normal limits
* No radiologic or clinical evidence of pancreatitis
* No history of organ transplant
* Patients with active infection requiring systemic treatment within 28 days prior to registration are not eligible
* Patients who are pregnant or nursing are not eligible; women of child bearing potential must have a negative serum or urine pregnancy test within 16 days prior to registration; women of child-bearing potential include:

  * Any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea >= 12 consecutive months)
  * Women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35m IU/mL
  * Women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy)
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2
* Archival tissue must be available for submission, though it is optional for patients to choose to participate in the correlative sub studies
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelet count >= 100,000/uL
* Hemoglobin >= 9 g/dL; patients may not have had a transfusion within 7 days prior to screening assessment
* Total bilirubin =< 1.5 x upper limits of normal
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN
* Albumin >= 2.8 g/dL
* Serum creatinine =< 1.5 x ULN, OR calculated creatinine clearance >= 30 mL/minute (modified Cockcroft and Gault formula)
* Urine protein to creatinine (UPC) ratio < 1.0; if UPC >= 1, then a 24-hour urine protein must be assessed; eligible patients must have a 24-hour urine protein value < 1 g
* Total serum calcium < 12 mg/dL
* International normalized ratio (INR) =< 1.2 x ULN; subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation
* TSH within normal limits (WNL); TSH only required for patients on thyroid supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2016-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni K Choueiri, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (488):
- United States (488):
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - San Diego VA Medical Center, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Montgomery Medical Center, Olney, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Veterans Administration, Columbia, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Hematology Oncology Associates of Central New York-Liverpool, Liverpool, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Hematology Oncology Associates of Central New York-Rome, Rome, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] George DJ, Hessel C, Halabi S, Michaelson MD, Hahn O, Walsh M, Picus J, Small EJ, Dakhil S, Feldman DR, Mangeshkar M, Scheffold C, Morris MJ, Choueiri TK. Cabozantinib Versus Sunitinib for Untreated Patients with Advanced Renal Cell Carcinoma of Intermediate or Poor Risk: Subgroup Analysis of the Alliance A031203 CABOSUN trial. Oncologist. 2019 Nov;24(11):1497-1501. doi: 10.1634/theoncologist.2019-0316. Epub 2019 Aug 9. PMID 31399500
- [Derived] Flaifel A, Xie W, Braun DA, Ficial M, Bakouny Z, Nassar AH, Jennings RB, Escudier B, George DJ, Motzer RJ, Morris MJ, Powles T, Wang E, Huang Y, Freeman GJ, Choueiri TK, Signoretti S. PD-L1 Expression and Clinical Outcomes to Cabozantinib, Everolimus, and Sunitinib in Patients with Metastatic Renal Cell Carcinoma: Analysis of the Randomized Clinical Trials METEOR and CABOSUN. Clin Cancer Res. 2019 Oct 15;25(20):6080-6088. doi: 10.1158/1078-0432.CCR-19-1135. Epub 2019 Aug 1. PMID 31371341
- [Derived] Choueiri TK, Hessel C, Halabi S, Sanford B, Michaelson MD, Hahn O, Walsh M, Olencki T, Picus J, Small EJ, Dakhil S, Feldman DR, Mangeshkar M, Scheffold C, George D, Morris MJ. Cabozantinib versus sunitinib as initial therapy for metastatic renal cell carcinoma of intermediate or poor risk (Alliance A031203 CABOSUN randomised trial): Progression-free survival by independent review and overall survival update. Eur J Cancer. 2018 May;94:115-125. doi: 10.1016/j.ejca.2018.02.012. Epub 2018 Mar 20. PMID 29550566
- [Derived] Choueiri TK, Halabi S, Morris MJ, George D. Reply to B. Rini et al and S. Buti et al. J Clin Oncol. 2017 Jun 1;35(16):1859-1860. doi: 10.1200/JCO.2017.72.2629. Epub 2017 Mar 6. No abstract available. PMID 28549224

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Cabozantinib-s-malate): Patients receive 60mg cabozantinib-s-malate PO QD for 6 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
- Arm II (Sunitinib Malate): Patients receive 50mg sunitinib malate PO QD for 4 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Sunitinib Malate)
Started | 79 | 78
Completed | 78 | 72
Not Completed | 1 | 6
Not completed — Withdrawal by Subject | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Sunitinib Malate) | Total
Number analyzed (Participants) | 79 | 78 | 157
Age, Continuous [Median (Full Range); unit: years] | 63 [40 to 82] | 64 [31 to 87] | 63 [31 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 21 | 34
  Male | 66 | 57 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 2 | 5
  White | 70 | 75 | 145
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) was investigator assessed and is measured from the beginning of treatment until patient progression or death. Progression was determined using RECIST 1.1 criteria, progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).The primary analysis will be based on the stratified log-rank statistic to compare the two treatment arms on PFS. The Kaplan-Meier product-limit estimator will be used to estimate PFS distributions.Progression Free Survival was assessed per investigator, as this was the protocol-specified endpoint, and both investigator and independent review analyses of the PFS endpoint have been published
Time Frame: Up to 5 years
Population: All patients that were enrolled on to study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Sunitinib Malate)
Number analyzed (Participants) | 79 | 78
Months | 8.2 [6.2 to 8.8] | 5.6 [3.4 to 8.1]
Statistical Analysis 1: Comparison: Arm I (Cabozantinib-s-malate) vs Arm II (Sunitinib Malate); Test type: Superiority; p = 0.012, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [.46 to .95]

2. Primary Outcome: Overall Survival (OS)
Description: The primary analysis will be based on the stratified log-rank statistic to compare the two treatment arms on OS. The Kaplan-Meier product-limit estimator will be used to estimate OS distributions.
Time Frame: Up to 5 years
Population: All enrolled patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Sunitinib Malate)
Number analyzed (Participants) | 79 | 78
Months | 30.3 [14.6 to 35.0] | 21.8 [16.3 to 27.0]
Statistical Analysis 1: Comparison: Arm I (Cabozantinib-s-malate) vs Arm II (Sunitinib Malate); Test type: Superiority; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.50 to 1.26]

3. Secondary Outcome: Objective Response Rates
Description: Objective response rates (ORR) was investigator assessed. ORR is the rate of complete or partial responses, based on RECIST 1.1 criteria. A response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. The Fisher exact test will be used to compare the two treatment arms.
Time Frame: Up to 5 years
Population: All enrolled patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Sunitinib Malate)
Number analyzed (Participants) | 79 | 78
proportion of participants | 0.33 [0.23 to 0.44] | 0.12 [0.054 to 0.21]

ADVERSE EVENTS:
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Sunitinib Malate)
Serious Adverse Events (participants affected / at risk) | 39/78 | 39/72
Other Adverse Events (participants affected / at risk) | 76/78 | 68/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cabozantinib-s-malate) (N=78) | Arm II (Sunitinib Malate) (N=72)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 5 (6)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (5)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5)
Death NOS (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 5 (6)
Fever (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 2 (2) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
ECG QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 3 (3)
Serum amylase increased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (3) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 8 (9) | 3 (3)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Thromboembolic event (Vascular disorders) | 7 (7) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cabozantinib-s-malate) (N=78) | Arm II (Sunitinib Malate) (N=72)
Anemia (Blood and lymphatic system disorders) | 29 (94) | 32 (103)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (7) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (2) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (3) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (1)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (5) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 4 (12) | 2 (3)
Hypothyroidism (Endocrine disorders) | 19 (50) | 4 (12)
Blurred vision (Eye disorders) | 2 (2) | 2 (3)
Dry eye (Eye disorders) | 1 (1) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (2)
Glaucoma (Eye disorders) | 1 (4) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (27) | 8 (12)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Bloating (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 16 (29) | 11 (15)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 54 (305) | 38 (96)
Dry mouth (Gastrointestinal disorders) | 16 (69) | 9 (14)
Dyspepsia (Gastrointestinal disorders) | 22 (56) | 12 (23)
Dysphagia (Gastrointestinal disorders) | 5 (8) | 2 (3)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 2 (18) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (26) | 4 (6)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (23) | 6 (10)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 6 (9) | 6 (15)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (3) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 30 (63) | 21 (50)
Nausea (Gastrointestinal disorders) | 25 (77) | 26 (40)
Oral dysesthesia (Gastrointestinal disorders) | 4 (14) | 2 (14)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 9 (12) | 5 (6)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 3 (4) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (29) | 14 (21)
Chills (General disorders) | 1 (1) | 4 (4)
Edema face (General disorders) | 2 (4) | 1 (3)
Edema limbs (General disorders) | 7 (38) | 10 (17)
Facial pain (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 65 (414) | 58 (215)
Fever (General disorders) | 3 (3) | 1 (1)
Flu like symptoms (General disorders) | 4 (4) | 3 (4)
Gait disturbance (General disorders) | 1 (3) | 1 (3)
Gen disord and admin site conds-Oth spec (General disorders) | 3 (5) | 5 (6)
Localized edema (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 8 (11) | 5 (12)
Sudden death NOS (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (3) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Corneal infection (Infections and infestations) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 5 (6) | 5 (6)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 4 (5)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (3) | 1 (1)
Skin infection (Infections and infestations) | 4 (6) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 4 (12) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (5) | 0 (0)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Activated partial throm time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 43 (135) | 19 (32)
Alkaline phosphatase increased (Investigations) | 10 (17) | 8 (10)
Aspartate aminotransferase increased (Investigations) | 49 (192) | 23 (36)
Blood bilirubin increased (Investigations) | 11 (18) | 4 (8)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
CPK increased (Investigations) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 2 (6) | 0 (0)
Creatinine increased (Investigations) | 18 (100) | 16 (55)
ECG QT corrected interval prolonged (Investigations) | 4 (6) | 5 (5)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 2 (7) | 1 (1)
Investigations - Other, specify (Investigations) | 7 (22) | 2 (2)
Lipase increased (Investigations) | 2 (6) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (24) | 14 (24)
Neutrophil count decreased (Investigations) | 12 (35) | 23 (93)
Platelet count decreased (Investigations) | 32 (131) | 43 (103)
Serum amylase increased (Investigations) | 2 (6) | 0 (0)
Weight gain (Investigations) | 0 (0) | 2 (3)
Weight loss (Investigations) | 28 (145) | 12 (32)
White blood cell decreased (Investigations) | 10 (39) | 24 (86)
Anorexia (Metabolism and nutrition disorders) | 37 (92) | 23 (46)
Dehydration (Metabolism and nutrition disorders) | 7 (10) | 6 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (30) | 11 (47)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (11) | 7 (9)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (47) | 13 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 16 (62) | 10 (14)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 13 (35) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 19 (92) | 8 (20)
Hyponatremia (Metabolism and nutrition disorders) | 12 (25) | 15 (24)
Hypophosphatemia (Metabolism and nutrition disorders) | 19 (62) | 11 (21)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 3 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (26) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (20) | 5 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (16) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (7) | 7 (9)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (8) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (16) | 2 (4)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 4 (33) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (52) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (16) | 6 (9)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 17 (32) | 15 (21)
Dysgeusia (Nervous system disorders) | 32 (98) | 21 (58)
Dysphasia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 9 (22) | 9 (16)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (8) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 3 (4) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 4 (14) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (6) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (41) | 4 (4)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 7 (13) | 3 (4)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 4 (8) | 4 (7)
Insomnia (Psychiatric disorders) | 8 (13) | 6 (11)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (11) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (18) | 4 (13)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (2)
Hematuria (Renal and urinary disorders) | 2 (4) | 2 (5)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 6 (14) | 9 (12)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (3) | 1 (4)
Urinary frequency (Renal and urinary disorders) | 2 (18) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (4) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (4) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (17) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (33) | 12 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 11 (32) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (19) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 8 (19) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (42) | 2 (6)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 16 (50) | 7 (8)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 33 (119) | 24 (100)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (16) | 4 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 12 (27) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 (26) | 9 (19)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 16 (71) | 8 (17)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (3)
Surgical and medical proced - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (11) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 64 (328) | 49 (193)
Hypotension (Vascular disorders) | 5 (5) | 2 (2)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less